CLINICAL TRIAL: NCT05520775
Title: Human Laboratory Screening of Semaglutide for Alcohol Use Disorder
Brief Title: Semaglutide for Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21-1689; R21AA026931-02 (NIH)
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Use Disorder; Cigarette Smoking
MeSH Terms: conditions — Alcoholism; Cigarette Smoking | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Randomized parallel group design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Participants will receive semaglutide via subcutaneous injections at escalating doses (.25mg to 1.0mg) over 9 weeks.
  Interventions: Drug: Semaglutide
- Sham/Placebo (Sham Comparator): Participants will receive sham subcutaneous injections over 9 weeks.
  Interventions: Drug: Sham/placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide (subcutaneous)
  Arms: Semaglutide
Drug: Sham/placebo — Sham subcutaneous injection
  Arms: Sham/Placebo

SUMMARY:
This is an early-Phase II human laboratory trial using a randomized, placebo-controlled, dose-ranging design to investigate the effects of semaglutide, a GLP-1 receptor agonist, on alcohol-related outcomes in adults with alcohol use disorder (AUD).

DETAILED DESCRIPTION:
This is an early-Phase II human laboratory trial using a randomized, placebo-controlled, dose-ranging design to investigate the effects of semaglutide, a GLP-1 receptor agonist, on laboratory alcohol responses and consumption, naturalistic alcohol consumption, and weight loss in participants with alcohol use disorder (AUD). Participants will attend weekly visits while semaglutide dosage is increased to 1.0mg over a period of approximately 9-10 weeks. Participants will attend weekly visits for medication or placebo administration. At scheduled intervals, participants will complete 4 laboratory sessions involving alcohol self-administration and alcohol challenge to characterize medication effects on alcohol-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* Meeting DSM-5 criteria for current (past year) alcohol use disorder (with 2-7 symptoms endorsed) and National Institute on Alcohol Abuse and Alcoholism (NIAAA) criteria for current at-risk drinking (i.e., >7/14 drinks in one week for women/men, with at least two episodes of 4+/5+ drinks in the past 30 days)
* Willingness/availability to take study medication and complete study procedures, including attending weekly visits for medication administration, side effect assessments, and glucose monitoring
* Willingness to complete laboratory sessions involving alcohol administration
* Ability to communicate and read in English

Exclusion Criteria:

* Reporting past 30-day use of illicit drugs other than cannabis at baseline, or having a positive toxicology screen for illicit drugs other than cannabis at baseline
* Meeting past-year criteria for a substance use disorder (with the exception of alcohol, tobacco or mild cannabis use disorder)
* Current engagement in alcohol treatments, or currently engaged in intentional efforts to quit alcohol use
* Past 30-day use of: Sincalide, Sulfonylureas, insulin and insulin products or other medications that may interact with semaglutide;, or weight control medications
* Prior use of semaglutide or other GLP-1 agonists
* Known or suspected hypersensitivity to study medication or related products
* Lifetime diagnosis of severe mental illness (including schizophrenia and bipolar disorder)
* History of suicide attempt, or recent (past 30 day) suicidal ideation, or psychiatric hospitalization in the last 6 months
* Current significant medical or neurological illness (based on self-report or medical record) including severe hepatic impairment or cirrhosis, impaired renal function (eGFR <50ml/min), acute or chronic pancreatitis, gastroparesis, gallbladder disease or cholelithiasis, other severe gastrointestinal disease, heart failure, coronary artery disease, stroke, seizure disorder, or other medical condition that poses a risk for the medication or alcohol administration components of the study (as determined by the MD)
* A personal or family history of medullary thyroid cancer or multiple endocrine neoplasia 2A or 2B
* Calcitonin greater than or equal to 50 ng/L
* Uncontrolled thyroid disease at screening
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g., subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* History of Type 1 or Type 2 diabetes, or HbA1c >6.5% measured at screening
* History of diabetic retinopathy, proliferative retinopathy, or maculopathy
* History of diabetic ketoacidosis
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and carcinoma in situ)
* Currently nursing, pregnant, anticipating pregnancy in the next 6 months, or not using a highly effective contraceptive method as judged by the MD, and defined as:

  1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  3. intrauterine device
  4. intrauterine hormone-releasing system
  5. bilateral tubal occlusion
  6. vasectomized partner
  7. sexual abstinence
* Elevation of serum lipase, amylase, direct (conjugated) bilirubin, or alkaline phosphatase (ALP), ALT, or AST) more than 3X the upper limit of normal on baseline bloodwork
* Baseline body mass index (BMI) <23kg/m^2
* Uncontrolled hypertension or systolic BP >180 mmHg and/or diastolic BP >105 mmHg, averaged from three measurements
* Plans for travel outside of the local area in the upcoming 12 weeks that would interfere with lab visits during the study period (or other logistic factors that would make it difficult to commit to entire duration of study)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hendershot, Ph.D., Principal Investigator — UNC-Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other investigators upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available following publication of study manuscripts and will be available indefinitely.
Access Criteria: Reasonable request from qualified investigator.

REFERENCES:
- [Derived] Hendershot CS, Bremmer MP, Paladino MB, Kostantinis G, Gilmore TA, Sullivan NR, Tow AC, Dermody SS, Prince MA, Jordan R, McKee SA, Fletcher PJ, Claus ED, Klein KR. Once-Weekly Semaglutide in Adults With Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Apr 1;82(4):395-405. doi: 10.1001/jamapsychiatry.2024.4789. PMID 39937469

RESULTS

PARTICIPANT FLOW:
Groups:
- Semaglutide: Participants will receive semaglutide via subcutaneous injections at escalating doses (0.25 mg to 1.0 mg) over 9 weeks.
  Semaglutide: Semaglutide (subcutaneous)
Period: Overall Study
Arm/Group | Semaglutide | Sham/Placebo
Started | 24 | 24
Completed | 23 | 19
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Sham/Placebo | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants] — Demographics Questionnaire
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 24 | 24 | 48
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — Demographics Questionnaire
  Years | 40.6 (10.5) | 39.0 (10.9) | 39.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 21 | 18 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Consumed
Description: Estimated grams of ethanol consumed.
Time Frame: Baseline (Week 0) to post-medication (Week 8)
Population: Participants who completed pre- and post-treatment laboratory self-administration.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 13 | 12
grams | -32.72 (27.98) | -6.95 (24.49)

2. Primary Outcome: Change in Breath Alcohol Concentration
Description: Peak breath alcohol concentration following an alcohol self-administration procedure.
Time Frame: Baseline (Week 0) to post-medication (Week 8)
Population: Participants who completed pre- and post-treatment laboratory self-administration.
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 13 | 12
g/dl | -0.034 (0.045) | -0.016 (0.047)

3. Secondary Outcome: Change in Subjective Stimulation (Biphasic Alcohol Effects Scale)
Description: Seven questions from the Biphasic Alcohol Effects Scale used to collect self-reported feelings of stimulation during an alcohol challenge procedure. Possible responses are 0-10, 0 being "not at all" and 10 being "extremely". Scale score ranges from 0 to 70. Higher scores indicate greater stimulation effects.
Time Frame: Baseline (Week 0) to post-treatment (Week 8)
Population: Participants with pre- and post-treatment data from an alcohol challenge laboratory session.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 22 | 18
Score on a scale | .45 (12.82) | -1.28 (13.49)

4. Secondary Outcome: Change in Subjective Sedation (Biphasic Alcohol Effects Scale)
Description: Seven questions from the Biphasic Alcohol Effects Scale used to collect self-reported sedative effects during an alcohol challenge procedure. Possible responses are 0 "not at all" through 10 "extremely". Scale scores range from 0 to 70. Higher scores indicate greater sedative effects.
Time Frame: baseline (Week 0) to post-medication (Week 8)
Population: Participants with pre- and post-treatment data from an alcohol challenge laboratory session.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 22 | 18
Score on a scale | 0.14 (10.69) | -3.22 (7.89)

5. Secondary Outcome: Change in Alcohol Demand (Alcohol Purchase Task)
Description: The Alcohol Purchase Task is a 20-question self-report measure which asks participants about the number of drinks they would purchase and consume based at different monetary costs. Intensity scores reflect the number of drinks that would be purchased when cost is zero.
Time Frame: Baseline (Week 0) to post-treatment (Week 8)
Population: Participants with pre- and post-treatment alcohol demand data.
Measure: Mean (Standard Deviation); unit: number of drinks
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 23 | 20
number of drinks | -2.91 (3.73) | -2.90 (7.82)

6. Secondary Outcome: Change in Cigarette Demand (Cigarette Purchase Task)
Description: Self-report cigarette demand as measured by the Cigarette Purchase Task. Intensity scores reflect the number of cigarettes that would be purchased when cost is zero.
Time Frame: Baseline (Week 0) to Post-medication (Week 8)
Population: Participants who reported cigarette use at baseline and provided pre- and post-treatment cigarette demand data.
Measure: Mean (Standard Deviation); unit: number of cigarettes
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 5 | 4
number of cigarettes | -2.4 (2.61) | -1.20 (2.17)

7. Secondary Outcome: Change in Daily Alcohol Use
Description: Self-reported drinks per day averaged across study week.
Time Frame: baseline (Week 0) to study endpoint (Week 10)
Population: Participants who have pre- and post- treatment data.
Measure: Mean (Standard Deviation); unit: daily drinks
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 21 | 18
daily drinks | -1.43 (1.51) | -0.81 (2.45)

8. Secondary Outcome: Change in Daily Cigarette Use
Description: Self-reported cigarettes per day
Time Frame: baseline (Week 0) to study endpoint (Week 10)
Population: Participants who reported cigarette use at baseline and have pre- and post-treatment data.
Measure: Mean (Standard Deviation); unit: daily cigarettes
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 5 | 4
daily cigarettes | -2.48 (4.22) | -1.30 (2.10)

9. Other Pre Specified Outcome: Change in Weight
Description: Change in Body weight
Time Frame: baseline (Week 0) to study endpoint (Week 10)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in HbA1c
Description: Hemoglobin A1C (HbA1c)
Time Frame: baseline (Week 0) to study endpoint (Week 10)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Alcohol Elimination
Description: Rate of alcohol elimination following an alcohol challenge procedure
Time Frame: baseline (Week 0) to post-medication (Week 8)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the Baseline medical visit through follow-up, a total of up to 12 weeks.
Arm/Group | Semaglutide | Sham/Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 22/24 | 18/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Semaglutide (N=24) | Sham/Placebo (N=24)
Decreased Appetite (Nervous system disorders) | 18 | 10
Nausea (Gastrointestinal disorders) | 17 | 4
Constipation (Gastrointestinal disorders) | 12 | 2
Headache (Nervous system disorders) | 12 | 5
Diarrhea (Gastrointestinal disorders) | 10 | 9
Fatigue (Nervous system disorders) | 9 | 6
Abdominal Pain (Gastrointestinal disorders) | 6 | 4
Dizziness (Nervous system disorders) | 3 | 2
Insomnia (Nervous system disorders) | 3 | 5
Increased Appetite (Nervous system disorders) | 2 | 4
Nervousness/Anxiety (Nervous system disorders) | 2 | 7
Vomiting (Gastrointestinal disorders) | 2 | 3
Depression (Psychiatric disorders) | 1 | 2
Increased Libido (General disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT05520775/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT05520775/ICF_003.pdf